CLINICAL TRIAL: NCT01580085
Title: Obstructive Sleep Apnea is Prevalent in Patients With Pulmonary Embolism
Brief Title: Obstructive Sleep Apnea in Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, meral uyar, Asisstant Professor, University of Gaziantep
Other Study IDs: gantep gogus 1
Record Dates: First submitted 2012-04-16; First posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Pulmonary Thromboembolism; Obstructive Sleep Apnea
Keywords: Sleep disordered breathing; gender; hypercoagulability
MeSH Terms: conditions — Pulmonary Embolism; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Coitus; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary embolism: Patients who were diagnosed with pulmonary embolism
  Interventions: Other: polysomnography
- control group: age and sex matched adults with osa and no thromboembolism
  Interventions: Other: polysomnography

INTERVENTIONS:
Other: polysomnography — full night supervised laboratory polysomnography
  Other Names: PSG

SUMMARY:
Obstructive sleep apnea (OSA) is a clinical syndrome characterized by repetitive closure of the airway and frequent awakenings during sleep. Repeated episodes of hypoxia, decrease in intrathoracic pressure, increased venous return and venous stasis, damage to vascular wall may ensue. An increased tendency for coagulation has also been reported in OSA. Venous stasis, vascular endothelial activation and hypercoagulability are also known risk factors for thromboembolism. All of these pathophysiologic changes in OSA may predispose patients for the development of pulmonary embolism (PE) however there is limited data about role of thromboembolic events in OSA.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients diagnosed with pulmonary embolism

Exclusion Criteria:

* less than 18 years of age
* any restrictive or obstructive lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects admitted to Department of Pulmonary Medicine of Gaziantep University who were diagnosed to have PE were included in the study group. Control group consisted of age and sex matched subjects without a clinic consistent with PE referred to the Sleep Clinic. PE was diagnosed when one or more of the following was present: compatible physical examination findings and multislice CT angiography or presence of deep venous thrombus (DVT) in addition to high risk with Wells criteria [5]. Subjects with any restrictive/obstructive lung pathology or younger than 18 years old were excluded.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meral Uyar, Assist Prof, Principal Investigator — University of Gaziantep
Locations (1):
- University of Gaziantep Hospital, Gaziantep, Turkey (Türkiye)